CLINICAL TRIAL: NCT03175302
Title: PREsurgical Cognitive Evaluation Via Digital clockfacEdrawing
Acronym: PRECEDE
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201700747-N; R01AG055337 (NIH); OCR18881 (Other: University of Florida)
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Cognitive Dysfunction
Keywords: cognitive processes; perioperative cognition; neurocognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical group: Baseline preoperative digital cognitive testing performance in adults to predict frequency and severity of clinician reported outcomes within the first three months post-surgery.
  Interventions: Behavioral: digital cognitive testing
- Control: Non-surgery matched peers with the same testing.
  Interventions: Behavioral: digital cognitive testing

INTERVENTIONS:
Behavioral: digital cognitive testing — The digital testing is hypothesized to identify latent features for differentiating cognitively impaired presurgical patient subgroups

SUMMARY:
This study leverages a modernized digital version of a well-known cognitive screening tool to examine pre and post operative cognitive function after surgery in adults age 65 years or more. Machine learning algorithms will be applied to the hospital wide standard of care cognitive metric to identify risk for post-operative cognitive complications.

DETAILED DESCRIPTION:
This proposal innovatively leverages a brief but informative digital test with machine learning to examine the subtlety of pre-surgery cognition within an extremely large number of older individuals screened preoperatively within an academic tertiary medical center. It also incorporates a unique group of well characterized non-surgery peers for demographic matching to assist with normal versus abnormal machine learning analyses.

ELIGIBILITY:
Inclusion Criteria:

* >/= 65 years of age
* screening within the University of Florida (UF) Health Preoperative clinic
* presurgical cognitive screening with the digital Clock Drawing Tool (dCDT)

Exclusion Criteria:

* < 65 years of age
* did not complete screening within the UF Health Preoperative clinic
* did not complete the presurgical cognitive screening with the digital Clock Drawing Tool (dCDT)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients >/= 65 years of age scheduled for screening within the UF Health Preoperative clinic
Sampling Method: Non-Probability Sample
Enrollment: 25240 (Estimated)
Dates: Start 2018-06-28 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Control and pre-surgery differences between digital behaviors | up to one year
  Measure range of digital outcome differences

SECONDARY OUTCOMES:
Predictive validity of digital behaviors on outcome | up to 1 year
  Digital tools will predict clinician reported events
Change over time in digital behavior between groups | up to 6-weeks
  Surgery group and control group differences from baseline to 6-weeks
Change over time in digital behavior between groups | up to 3-months
  Surgery group and control group differences from baseline to 3-months
Change over time in digital behavior between groups | up to one year
  Surgery group and control group differences from baseline to one year

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Price, Ph.D., Principal Investigator — University of Florida; Patrick Tighe, MD, MS, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bandyopadhyay S, Wittmayer J, Libon DJ, Tighe P, Price C, Rashidi P. Explainable semi-supervised deep learning shows that dementia is associated with small, avocado-shaped clocks with irregularly placed hands. Sci Rep. 2023 May 6;13(1):7384. doi: 10.1038/s41598-023-34518-9. PMID 37149670
- [Derived] Bandyopadhyay S, Dion C, Libon DJ, Price C, Tighe P, Rashidi P. Variational autoencoder provides proof of concept that compressing CDT to extremely low-dimensional space retains its ability of distinguishing dementia. Sci Rep. 2022 May 14;12(1):7992. doi: 10.1038/s41598-022-12024-8. PMID 35568709